CLINICAL TRIAL: NCT00003340
Title: A Phase II Study of Cyclophosphamide Followed by Topotecan in Patients With Refractory or Relapsed Acute Myelogenous Leukemia
Brief Title: Cyclophosphamide Plus Topotecan in Treating Patients With Refractory or Relapsed Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: J9736 CDR0000066314; JHOC-97100102; J-9736; NCI-G98-1435
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; Topotecan

INTERVENTIONS:
Drug: cyclophosphamide
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of cyclophosphamide plus topotecan in treating patients who have refractory or relapsed acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of cyclophosphamide followed by topotecan in patients with relapsed or refractory acute myelogenous leukemia. II. Confirm safety and tolerability of this combination on this schedule in these patients.

OUTLINE: Patients receive cyclophosphamide intravenously over 1 hour on day 1 followed by topotecan as a continuous 120 hour infusion starting 12 hours after completion of cyclophosphamide. Treatment may be repeated every 3-6 weeks for at least 2 courses.

PROJECTED ACCRUAL: A total of 26 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven acute myelogenous leukemia by bone marrow aspirate or biopsy Clear evidence of relapse or residual disease with greater than 5% blasts on bone marrow examination or greater than 30% peripheral blasts No active CNS leukemia Not eligible for potentially curative allogeneic or autologous bone marrow transplantation without further surgery Must have failed to achieve a complete remission with conventional chemotherapy (cytarabine based) or have relapsed within 12 months after initial remission

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 6 weeks Hematopoietic: See Disease Characteristics Hepatic: Bilirubin less than 1.6 mg/dL (unless due to disease) Renal: Creatinine less than 1.6 mg/dL (unless due to disease) No prior hemorrhagic cystitis Other: Not pregnant Fertile patients must use effective contraception No active uncontrolled infection

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics Recovered from prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: Must have recovered from prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-11; Primary Completion 2000-02 (Actual); Study Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Miller, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States